CLINICAL TRIAL: NCT03331445
Title: An Open Label Safety Study of Inhaled Gaseous Nitric Oxide (gNO) for Adults & Adolescents With Non-Tuberculous Mycobacteria, Burkholderia Spp, Aspergillus Spp and Corona-like Viral (Sub-Study) Infections
Brief Title: Inhaled Gaseous Nitric Oxide (gNO) Antimicrobial Treatment of Difficult Bacterial and Viral Lung (COVID-19) Infections
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid Incidence too low and Funding Completed
Sponsor: Chris Miller (Industry)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Chris Miller, CSO, Nitric Solutions Inc.
Organization: Nitric Solutions Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTM-CTP-01: H17-02107
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Tract Infections; Corona Virus Infection
Keywords: inhaled nitric oxide; non tuberculous mycobacteria; drug resistant pneumonia; Burkholderia; Aspergillus; COVID-19; Viral Envelope Proteins; SARS-COV-2
MeSH Terms: conditions — Respiratory Tract Infections; Coronavirus Infections; COVID-19 | interventions — Nitric Oxide; Nitrogen; Gases; Inhalation

STUDY DESIGN:
Intervention Model Description: Open label safety study (COVID-19 Sub-study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 160 ppm Nitric Oxide (Experimental)
  Interventions: Drug: Nitric Oxide 0.5 % / Nitrogen 99.5 % Gas for Inhalation

INTERVENTIONS:
Drug: Nitric Oxide 0.5 % / Nitrogen 99.5 % Gas for Inhalation — Inhaled Nitric Oxide 160ppm balance air
  Other Names: Thiolanox

SUMMARY:
Non tuberculous mycobacteria (NTM), Burkholdria spp, Aspergillus in the lung are almost impossible to eradicate with conventional antibiotics. In addition COVID-19 has know current treatment. These patients have few options to treat their lung infection. Nitric oxide has broad bactericidal and virucidal properties. It has been shown that nitric oxide was safe to be inhaled for similar cystic fibrosis patients and reduced drug resistant bacteria in the lungs. Further, research indicates that clinical isolates of NTM, Burkholderia spp, Aspergillus spp and Corona-like viruses can be eradicated by 160ppm NO exposure in the laboratory petri dish. This is not the first time inhaled NO treatment has been used in patients with difficult lung infections. This study will provide more data to see if NO therapy can reduce the bacterial load in the lungs, help the patients breath better; and in the case of COVID-19 act as a anti-viral agent resulting in the reduction of incidence of oxygen therapy, mechanical assistance of BIPAP, CPAP, intubation and mechanical ventilation during the study period.

DETAILED DESCRIPTION:
Main Study

Primary Objective: Assess the safety of inhaled NO (gNO) in adults & adolescents with NTM, Burkholderia, Aspergillus Lung Infections and Viral Lung (COVID-19) Infections

Safety will be evaluated by unanticipated adverse events in clinical labs (hematology, coagulation, and serum chemistries); in vitals; in inspired concentration of NO, O2 and NO2 delivered to each subject and; in real time methemoglobin and oxygen saturation levels.

Primary Endpoint:

Determine the safety of gNO in the NTM population,

* as confirmed by no unanticipated adverse events
* Absence of a deleterious mean change in FEV1% predicted (absolute) from baseline

Secondary safety Endpoint: Determine the efficacy of inhaled NO in adults with NTM, Burkholderia and Aspergillus Lung Infections

Efficacy will be evaluated by measuring the change in lung function with spirometry (specifically absolute change in FEV1 % predicted) from baseline to Days 5, 12, 19 and 26.

Secondary Efficacy Endpoint Determine the presence of an efficacy signal of gNO in the NTM, Burkholderia and Aspergillus Lung Infections

Efficacy will be assessed by the antimicrobial effect of inhaled NO on the density of NTM species and other microorganisms in sputum. Serial measurements of these microbial colony counts in sputum have been previously used as a measure of antimicrobial activity in other clinical trials of antibiotics in NTM.

• as confirmed by an improvement in pre-treatment bacterial colonization and post-treatment bacterial colonization on Days 19 and 26 as compared to baseline.

Efficacy will be assessed by change in Quality of Life Score.

* as assessed by an improvement in CRISS Score on Day 5, 19 and 26 as compared to baseline measurement;
* as determined by improvement in six-minute walk test with one minute recovery as compared to baseline measurement.

COVID-19 Substudy

Primary Endpoint:

Efficacy will be evaluated by measuring reduction in the incidence of mechanical assistance of BIPAP, CPAP, intubation and mechanical ventilation during the study period.

Secondary Endpoints:

1. Proportion of patients with mild COVID2019 who deteriorate to a severe form of the disease requiring mechanical intervention like BIPAP/CPAP, intubation and mechanical ventilation;
2. Mortality from all causes during the study period;
3. Negative conversion of COVID-19 RT-PCR from upper respiratory tract measured as the proportion of patients with a negative conversion of RT-PCR from an oropharyngeal or a nasopahryngeal swab;
4. Time to clinical recovery defined as the time from initiation of the study to discharge or to normalization of fever (defined as <36.6°C from axillary site, or < 37.2°C from oral site or < 37.8°C from rectal or tympanic site), respiratory rate (< 24 bpm while breathing room air);
5. Alleviation of symptoms recorded in the Modified Jackson Cols score with particular definition of cough (defined as mild or absent in a patient reported scale of severity).

ELIGIBILITY:
COVID SubStudy Inclusion Criteria

* Capable of understanding and providing signed informed consent and ability to adhere to the requirements and restrictions of this protocol;
* Men and Women ≥ 19 years of age unless local laws dictate otherwise;
* English speaking;
* Suspected of exposure to SARS-CoV-2 with fatigue and at least a fever (>37.90 C) or cough or sore throat or a positive swab for SAR-CoV-2 within 5 days of the of enrollment;
* Must be willing to use an adequate form of contraception (or abstinence) from the time of the first dose with the IMP until after the last dose of IMP.

Exclusion Criteria

* Prior Tracheostomy;
* Concomitant treatment involving high flow nasal cannula;
* Any clinical contraindications, as judged by the attending physician;
* Mentally or neurologically disabled patients who are considered not fit to consent to their participation in the study;
* Prior COVID-19 infection or a positive swab for SARS-CoV-2 greater than 5 days from enrollment;
* Family members in the same household already on the study;
* Hydroxychloroquine, colchicine and other experimental antiviral medications;
* unwilling to practice a medically acceptable form of contraception from screening to Day 26 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent).

Recruitment on hold for following Criteria during COVID-19 Pandemic

Inclusion Criteria:

* Written informed consent.
* Has been previously diagnosed with NTM, Burkholderia spp and Aspergillus spp. or Corona-like viral infection:

  1. NTM, Burkholderia spp and Aspergillus spp defined as positive culture(s) of at least one species of Mycobacterium avium Complex (MAC) or Mycobacterium abscessus Complex (MABSCor Burkholderia spp and Aspergillus spp) or Corona-like viral infection:
  2. History of repeatedly positive cultures (2 or more), irregardless of therapy
* Male or female ≥14 years of age.
* Female not pregnant at time of study.
* Has an FEV1 ≥ 30 % of predicted. c. Suspected corona-like viral infection
* Oxygen saturation on room air >92% at screening.

  a. Able to breathe without supplemental oxygen for 60 minutes
* Non-smoker for at least 6 months prior to screening and agrees not to smoke during the study.
* Willing and able to comply with the treatment schedule and procedures.

Exclusion Criteria:

* Use of an investigational drug within 30 days of screening
* History of frequent epistaxis (>1 episode/month)
* Significant hemoptysis within 30 days (≥ 5 mL of blood in one coughing episode or > 30 mL of blood in a 24 hour period)
* History of reactive pulmonary vascular hypertension
* Methemoglobin >3% at screening
* Liver function insufficiency (ALT/ AST >3 of normal values)
* Hemoglobin <11 g/dl
* Thrombocytopenia (platelet count <100,000/mm3) at screening
* Prothrombin time international ratio (INR) > 1.3 at screening
* Changes to antibiotics (e.g. azithromycin) from 7 days prior to screening through last treatment day. (Subjects may be taking antibiotics or antivirals during this time period, but they cannot start, stop or change doses during this time period)
* On supplemental oxygen during gNO treatment (SaO2 < 90% for 50 minutes while resting in a chair).
* For women of child bearing potential:

  1. positive pregnancy test at screening or
  2. lactating or
  3. unwilling to practice a medically acceptable form of contraception from screening to Day 36 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent)
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Measure the safety of 160ppm inhaled nitric oxide delivery in NTM subjects | 26 Days
  Measure the number of unanticipated adverse events over the duration of the study protocol

SECONDARY OUTCOMES:
Measure the effect of 160ppm inhaled nitric oxide delivery on lung spirometry in NTM subjects | Day 5,12,19 and 26
  Measure the change in absolute FEV1.0 change from baseline during 160 ppm inhalation therapy
Measure the antimicrobial effect of 160ppm inhaled nitric oxide on lung NTM bacterial load in the sputum | Day 19 and 26
  Measure the difference from baseline NTM species bacterial load (0 to +4) in sputum during 160ppm nitric oxide inhalation therapy
Measure the effect of 160ppm inhaled nitric oxide on Quality of Life (CRISS) Score | Day 19 and 26
  Measure the difference from baseline CRISS (0-100) during 160ppm nitric oxide inhalation therapy (lower score represents higher quality of life)

OTHER OUTCOMES:
Sub-Study Primary Endpoint(s): Efficacy to reduce respiratory interventions | Day 26
  Measuring reduction in the incidence of mechanical assistance including oxygen therapy, BIPAP, CPAP, intubation and mechanical ventilation during the study period.
Efficacy in reduction of mortality | Day 26
  Measured by death from all causes
Antiviral effect | Day 26
  Assessed by time to negative conversion of COVID-19 RT-PCR from upper respiratory tract
Efficacy on clinical improvement | Day 26
  Time to clinical recovery as measured by resolution of clinical signs
Efficacy on the respiratory symptoms | Day 26
  Measured by change in the Modified Jackson Cold Score

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Road, MD, Principal Investigator — MD
Locations (1):
- Nitric Solutions-Mobile Unit, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deppisch C, Herrmann G, Graepler-Mainka U, Wirtz H, Heyder S, Engel C, Marschal M, Miller CC, Riethmuller J. Gaseous nitric oxide to treat antibiotic resistant bacterial and fungal lung infections in patients with cystic fibrosis: a phase I clinical study. Infection. 2016 Aug;44(4):513-20. doi: 10.1007/s15010-016-0879-x. Epub 2016 Feb 9. PMID 26861246
- [Background] Miller C, Miller M, McMullin B, Regev G, Serghides L, Kain K, Road J, Av-Gay Y. A phase I clinical study of inhaled nitric oxide in healthy adults. J Cyst Fibros. 2012 Jul;11(4):324-31. doi: 10.1016/j.jcf.2012.01.003. Epub 2012 Apr 18. PMID 22520076
- [Background] Yaacoby-Bianu K, Gur M, Toukan Y, Nir V, Hakim F, Geffen Y, Bentur L. Compassionate Nitric Oxide Adjuvant Treatment of Persistent Mycobacterium Infection in Cystic Fibrosis Patients. Pediatr Infect Dis J. 2018 Apr;37(4):336-338. doi: 10.1097/INF.0000000000001780. PMID 28885458